CLINICAL TRIAL: NCT06920823
Title: Comparison of Antegrade and Retrograde Fixation With Intramedullary Headless Canulated Screws in Patients With Metacarpal Fractures
Brief Title: Comparison of Antegrade and Retrograde Fixation With Intramedullary Screws in Metacarpal Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, assistant professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111990
Record Dates: First submitted 2025-03-21; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Metacarpal Fracture
Keywords: Metacarpal Fracture, Intramedullary Fixation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): antegrade (proximal entry) fixation
  Interventions: Procedure: antegrade (proximal entry) fixation
- Group 2 (Active Comparator): retrograde (distal entry) fixation
  Interventions: Procedure: retrograde (distal entry) fixation

INTERVENTIONS:
Procedure: antegrade (proximal entry) fixation — In the antegrade headless cannulated screw fixation technique, a small incision was made on the extensor aspect of the fractured metacarpal at the level of the carpometacarpal joint.
  Arms: Group 1
Procedure: retrograde (distal entry) fixation — In the fixation technique with retrograde headless cannulated screw, a small incision was made on the extensor side of the fractured metacarpal at the level of the metacarpophalangeal joint.
  Arms: Group 2

SUMMARY:
Purpose: Intramedullary fixation has proven to be an efficacious intervention for metacarpal fractures. Advantages involve stable fixation facilitating early surgical rehabilitation and higher fracture union rates, without increased morbidity. We aimed to compare the results of fixation of metacarpal fractures with headless cannulated screws towards antegrade or retrograde on pain, function and quality of life in patients with metacarpal fractures.

Methods: Patients admitted to Pamukkale University Orthopedics and Traumatology Department, due to metacarpal fracture were prospectively included in the study and randomly grouped. A total of 22 patients and 26 metacarpal fractures were assessed. Group I patients were operated with antegrade(proximal entry) , and group II with retrograde (distal entry) , using intramedullary headless cannulated screws. Appropriate screw selection was made by measuring the metacarpal isthmus diameter of the patient's x-ray results (AP and oblique direction). We used headless cannulated screws with diameters between 3.5mm and 5mm in the fractures.

DETAILED DESCRIPTION:
This was a prospective randomised comparative single-blinded study comparing the effects of intramedullary fixation direction and entry site in patients with metacarpal fractures.

The participants were first evaluated at post-operative 6th week and the last evaluation was performed at post-operative 12th week The evaluations included radiographic union, grip strength measurement (with Jamar hydraulic hand dynamometer), range of motion measurement (compared to the opposite hand), and Michigan Hand Outcome Questionnaire (MHQ) questionnaire. All assessments were performed by the same investigator. The researcher who performed the evaluations did not know which group the participants were in.

In the antegrade headless cannulated screw fixation technique, a small incision was made on the extensor aspect of the fractured metacarpal at the level of the carpometacarpal (CMC) joint and the extensor tendon was excised. After fracture reduction, k-wire was inserted intramedullarly. After appropriate drilling, 1 headless cannulated screw was applied distally.(figure 1) In the fixation technique with retrograde headless cannulated screw, a small incision was made on the extensor side of the fractured metacarpal at the level of the MCP joint, and the extensor tendon split was passed. After fracture reduction, k-wire was inserted intramedullarly. After appropriate drilling, headless cannulated screw was applied proximally.

ELIGIBILITY:
Inclusion Criteria:

* Operated for metacarpal fracture,
* Speak and understand Turkish,
* Understand the verbal and written information given.
* Regular follow-up visits

Exclusion Criteria:

* Open epiphysis
* Pathological fractures
* Fractures requiring bone grafting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Radiographic Examination (anteroposterior and oblique diameter) | postop 6th week
  Primary bone healing was accepted as union when callus tissue developed in at least 3 cortices on AP and oblique radiographs taken with a radiography device or on the 6th week control radiograph. Radiological measurements were performed by a single observer.

SECONDARY OUTCOMES:
Range of motion | postop 6th and 12th week
  Range of motion was measured with a universal goniometer. All measurements were made with the patient in the sitting position.
Grip strength | postop 12th week
  Grip strength was assessed as gross grip and pinch grip with a Jamar hand dynamometer and a pinchmeter according to the recommendation by the American Society of Hand Therapists.
Hand functionality (Michigan Hand Outcomes Questionnaire) | postop 12th week
  Michigan Hand Outcomes Questionnaire consists of a total of 63 items for both hands and each item is scored between 1-5. It evaluates the hand and wrist in 6 domains: overall hand function, activities of daily living, pain, work performance, aesthetics, and patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Eraslan, PhD, Principal Investigator — Faculty of Physiotherapy and Rehabilitation
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No